CLINICAL TRIAL: NCT04888975
Title: A Non-randomized, Open-Label Study to Evaluate the Safety and Effectiveness of the Dayspring Technology for Patients With Breast Cancer Related Lymphedema (BCRL) After Lymphatic Surgery
Acronym: TIGRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCT 005
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Lymphedema; Lymphedema, Breast Cancer; Lymphedema Arm
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Breast-cancer related lymphedema (BCRL) after lymphatic surgery (Experimental): Patients with Breast-cancer related lymphedema (BCRL) after lymphatic surgery
  Interventions: Device: Dayspring Active Wearable Compression System

INTERVENTIONS:
Device: Dayspring Active Wearable Compression System — Dayspring Active Wearable Compression System

SUMMARY:
To evaluate the Dayspring Active Wearable Compression Technology in enhancing lymph movement and its safety and effectiveness after lymphatic surgery

DETAILED DESCRIPTION:
To evaluate the Dayspring Active Wearable Compression Technology in enhancing lymph movement and its safety and effectiveness after lymphatic surgery

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of upper extremity edema and have or will undergo lymphatic surgery with Dr. Nguyen
* Subjects must have a difference in volume greater than 3% between the limbs.

Exclusion Criteria:

* Individuals with a history or presence of a systemic disorder or condition that could place the patient at increased risk from sequential compression therapy
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Patients with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
* Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer
* Patients must not have any diagnosed cognitive or physical impairment that would interfere with use of the device
* Diagnosis of lipedema
* Diagnosis of acute infection. The source of the infection must be treated for 2 weeks prior to admittance into the study
* Diagnosis of acute thrombophlebitis (in last 2 months)
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled)
* Diagnosis of chronic kidney disease
* Diagnosis of epilepsy
* Patients with poorly controlled asthma
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days
* Bilateral limb edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ICG Fluorescence Lymphatic Imaging | Baseline and at Day 28
  ICG fluorescence lymphatic imaging evaluates for changes in lymphatic drainage of the limb. ICG is a water soluble tricarbocyanine dye, has a short plasma half life of 3 to 5 minutes in humans, is excreted exclusively by the liver into the bile, and is not associated with risk for nephrotoxicity. ICG contains sodium iodide and is recommended by manufacturer to be used with caution in patients who have a history of allergy to iodides, although type-I allergic reaction (anaphylaxis) cannot really occur because iodine is a chemical element that is an essential component of the human body.

CONTACTS AND LOCATIONS:
Locations (1):
- Dung Nguyen, MD, PharmD, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No